CLINICAL TRIAL: NCT04820439
Title: Pharmacokinetic Study of Recombinant Monoclonal Antibody Against Human Epidermal Growth Factor Receptor Injection (HS627) and Perjeta ® in Healthy Male Subjects: a Randomized, Double-blind, Parallelity-controlled Study
Brief Title: Pharmacokinetic Study of Recombinant Monoclonal Antibody Against Human Epidermal Growth Factor Receptor Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS627-BE
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- recombinant monoclonal antibody against human epidermal growth factor receptor injection (HS627) (Experimental)
  Interventions: Drug: recombinant monoclonal antibody against human epidermal growth factor receptor injection (HS627)
- Perjeta ® (Active Comparator)
  Interventions: Drug: Perjeta ®

INTERVENTIONS:
Drug: recombinant monoclonal antibody against human epidermal growth factor receptor injection (HS627) — A single intravenous infusion of HS627 420mg
  Arms: recombinant monoclonal antibody against human epidermal growth factor receptor injection (HS627)
Drug: Perjeta ® — A single intravenous infusion of Perjeta ®420mg
  Arms: Perjeta ®

SUMMARY:
This study was designed as a randomized, double-blind, parallelity-controlled study.Eighty-eight healthy male subjects (44 in each group) will be enrolled in this study.The aim of this clinical trial is to evaluate pharmacokinetic similarity between recombinant monoclonal antibody against human epidermal growth factor receptor injection (HS627) and Perjeta ® in a single intravenous infusion in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 18-40.
* The body mass index is in the range of 19-26 kg/m2 (including thecritical value). The weight is 50 kg-80kg.
* The subjects have no family planning within 3 months and could select contraceptive method
* The subjects who have signed the informed consent and are able to complete the experiment according to the trial protocol.
* Echocardiography showed left ventricular ejection fraction (LVEF) > 50% ,which two weeks before administration of experimental drug.

Exclusion Criteria:

* The subjects with a history of malignant tumor.
* The subjects who has received any live vaccine within 6 months prior to signing the informed consent.
* The subjects who has upper respiratory tract infection or other acute infections within the previous 2 weeks of screening.
* The subjects who had undergone surgery within 2 months prior to signing the informed consent.
* Anti-drug antibody (ADA) detection positive.
* Previous treatment with any antibody targeting the HER2 receptor or Those who have used monoclonal antibodies within 6 months prior to signing the informed consent.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC)0-∞ | 150 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞
Area under the plasma concentration versus time curve (AUC)0-t | 150 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Peak Plasma Concentration (Cmax) | 150 days
  Evaluation of Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
The total clearance(CL) | 150 days
  Evaluation of the total clearance(CL)
elimination half-life time(T1/2) | 150 days
  Evaluation of elimination half-life time(T1/2)

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China